CLINICAL TRIAL: NCT03275220
Title: Assessment Of Right Ventricular Function In Patients Undergoing Coronary Artery Bypass Graft In Assiut University
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mero Fouad, Principal Investigator, Assiut University
Other Study IDs: 17100309
Record Dates: First submitted 2017-08-27; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: CORONARY ARTERY BYPASS
MeSH Terms: interventions — Echocardiography; Echocardiography, Three-Dimensional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 2D Echocardiography and 3D Echocardiography — Imaging of right ventricle by 2d echocardiography and 3D echocardiography to assess right ventricular function accurately

SUMMARY:
Assessment Of Right Ventricular Function In Patients Undergoing Coronary Artery Bypass Graft In Assiut University

DETAILED DESCRIPTION:
Right ventricular (RV) dysfunction is a major risk factor in coronary artery disease (CAD) and patient undergoing revascularization with this combination , incidence of RV dysfunction is reported in about 20% cases of CAD.

RV dysfunction is a possible cause of cardiac failure after cardiac surgery and has a high mortality rate.

RV dysfunction is a recognized cause of hypotension early after coronary artery bypass graft surgery (CABG)

A decrease in RV function is an event known to occur after CABG. Right ventricular dysfunction can be seen during and immediately after cardiac surgery. Although the mechanism of this phenomenon is not well understood, cardiopulmonary bypass, perioperative myocardial ischemia, intraoperative myocardial damage, cardioplegia, and pericardial disruption or adhesion have been suggested as probable causes.

Major reasons for complications of cardiac surgery are the need for hypothermic cardiac arrest, aortic cross clamping, and exposure to a cardiopulmonary bypass circuit.

It has been postulated that avoidance of these factors by performing off-pump coronary artery bypass (OPCAB) surgery might reduce perioperative morbidity and improve outcome.

Recently, the portion of coronary artery bypass grafting on the beating heart without the use of cardiopulmonary bypass (CPB) has been expanded in cardiac surgery as a result of awareness of the damaging effect of CPB

Whether OPCAB surgery can fulfill these expectations, or to which degree, is yet unclear.

A few studies on hemodynamic alternations associated with OPCAB reported that reduced functions of both ventricles during coronary artery anastomosis are the main mechanism of hemodynamic derangements and especially, impaired diastolic function of the right ventricle (RV) plays an important role

However, clinical studies evaluating the change in RV function in patients with ischemic heart disease are very rare. It is reported that the major cause of hemodynamic changes during OPCAB was disturbed diastolic filling of the RV through the measurement of chamber pressures or monitoring of echocardiography.

There was no significant change in the RVEF and cardiac index during anastomosis of the left anterior descending artery and right coronary artery. However, the significantly reduced RVEF accompanied by an increase in RV afterload and decrease in the CO was observed during anastomosis of the obtuse marginal (OM) artery. RV volumes did not significantly change during anastomoses, though the right atrial pressure increased during anastomoses of all coronary arteries. The displacement of beating heart for positioning during anastomosis of the graft to OM artery caused significant derangement of RV function and decrease in CO.

ELIGIBILITY:
1. Inclusion criteria:

   • Patients will undergo elective CABG in Assiut university hospital
2. Exclusion criteria:

   * Poor echo window.
   * Refusal of the patient
   * Patients with prior RV dysfunction.
   * Patients with LV dysfunction (EF:<40%).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include patients will undergo elective CABG of different ages from cardiology department, Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-09-10 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of effects of CABG on right ventricular function | 6 months
  assessment of right ventricular function in patients undergoing CABG using 2D echocardiography and 3D echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Salah Atta, Study Chair — professor; Salma Taha, Study Chair — lecturer
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roshanali F, Yousefnia MA, Mandegar MH, Rayatzadeh H, Alinejad S. Decreased right ventricular function after coronary artery bypass grafting. Tex Heart Inst J. 2008;35(3):250-5. PMID 18941594